CLINICAL TRIAL: NCT05452187
Title: Evaluation of the Safety and Effectiveness of Direct-acting Antiviral Drugs in the Treatment of Hepatitis C in Patients With Inflammatory Bowel Disease: National Multicenter Study (MIC Project).
Brief Title: Evaluation of the Safety and Effectiveness of Direct-acting Antiviral Drugs in the Treatment of Hepatitis C in Patients With Inflammatory Bowel Disease: National Multicenter Study
Acronym: MIC project
Status: Completed | Type: Observational
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Other Study IDs: MIC2020
Record Dates: First submitted 2022-06-10; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Inflammatory Bowel Diseases; Hepatitis C Virus Infection
Keywords: Inflammatory Bowel Diseases; Hepatitis C Virus Infection; Direct-acting antiviral drugs
MeSH Terms: conditions — Inflammatory Bowel Diseases; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with IBD and chronic HCV infection treated with DAAs and/or interferon.: Cohort patients with IBD and chronic HCV infection treated with DAAs and/or interferon collected from the ENEIDA database.
  Interventions: Drug: Assess the effectiveness and safety of DAAs in patients with IBD.; Drug: Evaluate the interaction of DAAs with IBD drugs, particularly immunosuppressants and/or biologics.; Other: Assessment of the impact of DAAs on the course of IBD.

INTERVENTIONS:
Drug: Assess the effectiveness and safety of DAAs in patients with IBD. — Variables evaluated: age, gender, location, extent, phenotype, and activity of IBD, treatments, anti-HCV and viral load, DAA treatment and duration, fibrosis and hepatic decompensation and adverse effects (AE).
  Other Names: Direct-acting antiviral (DAA) to treat hepatitis C virus (HCV) infection in inflammatory bowel disease (IBD) patients.
Drug: Evaluate the interaction of DAAs with IBD drugs, particularly immunosuppressants and/or biologics. — Variables evaluated: Interactions.
Other: Assessment of the impact of DAAs on the course of IBD. — Qualitative variables will be expressed as a percentage and 95% confidence interval and quantitative variables as median and interquartile range. A priori it is difficult to determine which statistical analysis should be performed. It is basically a descriptive study, and the subsequent statistical analysis will depend on the evolution that the patients have presented in relation to the DAA treatment. If the drugs have been well tolerated without adverse effects, further statistical analysis will not be necessary. Instead, if the DAAs trigger activity outbreaks, variables related to the appearance of these outbreaks will be evaluated (type of DAA, immunomodulator, ...). To compare whether there are differences between the established groups, Chi Square (in qualitative independent variables), a t-student or ANOVA or their corresponding non-parametric tests (in quantitative independent variables) will be used. Statistical significance has been set at a probability level of <0.05.

SUMMARY:
The prevalence of hepatitis C virus infection (HCV) in patients with inflammatory bowel disease (IBD) ranges from 1-6%. Direct-acting antivirals (DAAs), with cure rates >90%, represent a radical change from interferon-based therapies. The ECCO (European Crohn's and Colitis Organisation) guidelines (Kucharzik T, Ellul P, Greuter T, et al. ECCO Guidelines on the Prevention, Diagnosis, and Management of Infections in Inflammatory Bowel Disease. J Crohn's Colitis. 2021;15(6):879-913) warns about the risk of IBD reactivation due to the effect of DAAs, but HCV management in this situation is uncertain given the lack of evidence.

The project is proposed as the largest retrospective multicenter descriptive study carried out to evaluate the use of DAAs for HCV eradication in patients with IBD. The Eneida database (Zabana Y, Panés J, Nos P, et al. The ENEIDA registry (Nationwide study on genetic and environmental determinants of inflammatory bowel disease) by GETECCU: Design, monitoring, and functions. Gastroenterol y Hepatol. 2020;43(9):551-8.) of the Spanish Working Group on Crohn's Disease and Ulcerative Colitis (GETECCU) is an adequate registry to identify patients with HCV infection. The serological status of the infection is frequently recorded in the ENEIDA database, and it is generally evaluated at the time of IBD diagnosis, before starting immunosuppressive treatment. The ENEIDA registry has the advantage over large population studies that researchers have access to relevant details of the clinical history, which can respond to the controversies raised.

This multicenter retrospective descriptive study will provide useful information to be able to give evidence-based recommendations regarding treatment of HCV in patients with IBD.

DETAILED DESCRIPTION:
Hypothesis:

The use of DAAs for HCV eradication in patients with IBD is effective and safe. DAAs do not trigger IBD flares. DAAs probably do not present serious pharmacological interactions, with clinically relevant, with immunosuppressants and/or biological agents.

ELIGIBILITY:
Inclusion Criteria:

* All individuals diagnosed with IBD according to the ECCO criteria and chronic HCV infection (positive HCV Ab and detectable RNA) treated with DAAs and/or interferon collected in the ENEIDA database, and who have properly completed the fields of age, gender, treatment, location, and phenotype of IBD, will be included in the study.
* Study period: Patients treated with DAAs between January 1, 2011 - February 28, 2021.

Exclusion Criteria:

* Spontaneous cure of HCV without treatment
* HCV treatment outside the study period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with HCV Ab (positive/negative) and with RNA (detectable/undetectable) will be identified using the ENEIDA database.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Percentage of sustained viral response (effectiveness) in patients with IBD and HCV infection treated with DAAs. | 8 weeks
Number and description of adverse events (safety) and possible interactions of DAAs with IBD drugs, particularly immunosuppressants and/or biologics. | 8 weeks

SECONDARY OUTCOMES:
Compare the clinical Crohn's disease activity (measured by Harvey Bradshaw Index) before and during the treatment with DAAs, to assess the impact of DAAs on the course of IBD. | 8 weeks
  Harvey Bradshaw Index (HBI) for Crohn's disease (CD): The minimum score obtainable is 0, which indicates the absence of disease. The maximum attainable score depends on the number of stools the patient identifies per day, however, it is in the range of 18.
  HBI score interpretation: < 5 remission, 5-7 points (mild activity), 8-16 points (moderate activity), > 16 points (severe activity).
Compare the clinical ulcerative colitis activity (measured by Partial Mayo Score) before and during the treatment with DAAs, to assess the impact of DAAs on the course of IBD. | 8 weeks
  Partial Mayo Score in ulcerative colitis (UC): The minimum score obtainable is 0, which indicates the absence of disease. The maximum attainable score is 9.
  Partial Mayo score interpretation: < 2 remission, 2-4 points (mild activity), 5-7 points (moderate activity), >7 points (severe activity).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Esteve, PhD, MD, Principal Investigator — Hospital Universitari Mútua Terrassa
Locations (1):
- Hospital Universitari Mutua Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kucharzik T, Ellul P, Greuter T, Rahier JF, Verstockt B, Abreu C, Albuquerque A, Allocca M, Esteve M, Farraye FA, Gordon H, Karmiris K, Kopylov U, Kirchgesner J, MacMahon E, Magro F, Maaser C, de Ridder L, Taxonera C, Toruner M, Tremblay L, Scharl M, Viget N, Zabana Y, Vavricka S. ECCO Guidelines on the Prevention, Diagnosis, and Management of Infections in Inflammatory Bowel Disease. J Crohns Colitis. 2021 Jun 22;15(6):879-913. doi: 10.1093/ecco-jcc/jjab052. No abstract available. PMID 33730753
- [Background] Zabana Y, Panes J, Nos P, Gomollon F, Esteve M, Garcia-Sanchez V, Gisbert JP, Barreiro-de-Acosta M, Domenech E; en representacion de GETECCU. The ENEIDA registry (Nationwide study on genetic and environmental determinants of inflammatory bowel disease) by GETECCU: Design, monitoring and functions. Gastroenterol Hepatol. 2020 Nov;43(9):551-558. doi: 10.1016/j.gastrohep.2020.05.007. Epub 2020 Jul 14. English, Spanish. PMID 32674882